CLINICAL TRIAL: NCT05126056
Title: Lipid Lowering Effect of Plant Stanol Ester in a Drinkable Non-dairy Product
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Raisio Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NGH2
Record Dates: First submitted 2021-11-09; First posted 2021-11-18 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-12

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — plant stanol ester

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Comparator (Active Comparator): Products that contain plant stanol ester. Product with active ingredient
  Interventions: Other: Plant stanol ester
- Placebo comparator (Placebo Comparator): Placebo product. Product without active ingredient
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Plant stanol ester — Product with active ingredient vs product without active ingredient
  Arms: Active Comparator
Other: Placebo — Placebo
  Arms: Placebo comparator

SUMMARY:
The aim is to determine the effect of investigational products on serum LDL cholesterol.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Mildly or moderately elevated plasma cholesterol levels (plasma total cholesterol 5.5-8.0 mmol/l)
* Plasma triglyceride levels ≤ 4.0 mmol/l
* Age 18-65 years

Exclusion Criteria:

* Intolerance to oats or other ingredients of the test products
* Severe obesity (BMI ≥ 32 kg/m2)
* Consumption of lipid/cholesterol lowering medication (e.g. ezetimibe, PCSK9 inhibitors, resins, fibrates) 1 month prior to the screening visit and throughout the study. Statin treatment is allowed at stable dose.
* Consumption of plant stanol or plant sterol containing food products or supplements or other foods or supplements such as beta-glucan enriched foods, red rice, berberine or any combination of these used for cholesterol lowering purpose 1 month prior the study entry (baseline blood sample)
* History of malignant diseases like cancer within five years prior to recruitment
* History of unstable coronary artery disease (myocardial infarction, coronary artery bypass graft (CABG), percutaneous transluminal coronary angioplasty (PTCA) within the previous 6 months
* Diagnosed type 1 or type 2 diabetes requiring medical treatment
* Celiac disease
* Medically prescribed diet/treatment for slimming or a special diet like very low calorie diet or use of prescribed an obesity drug (e.g. Orlistat, Victoza)
* Alcohol abuse (> 4 portion/per day) or recreational drug abuse
* Pregnancy or planned pregnancy or lactating
* Clinically significant abnormalities in screening labs
* Participation in another clinical trial in the preceding 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in low-density lipoprotein (LDL) cholesterol concentration (%) | 0 vs 3 weeks
  Mean relative change in serum LDL cholesterol concentration during the intervention

SECONDARY OUTCOMES:
LDL cholesterol concentration | 0 vs 3 weeks
  Mean absolute change in serum LDL cholesterol concentration during the intervention between test and control group
total cholesterol concentration | 0 vs 3 weeks
  Changes in serum total cholesterol concentration during the intervention
High density lipoprotein (HDL) cholesterol concentration | 0 vs 3 weeks
  Changes in serum HDL cholesterol concentration during the intervention
non-HDL cholesterol concentration | 0 vs 3 weeks
  Changes in serum non-HDL cholesterol concentration during the intervention
Total triglyceride concentration | 0 vs 3 weeks
  Changes in serum triglycerides concentrations
Nuclear magnetic resonance (NMR) blood biomarkers | 0 vs 3 weeks
  Changes in specific NMR blood biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Helena Gylling, Principal Investigator — Helsinki University Hospital, Helsinki, Finland
Locations (1):
- Nightingale Health plc, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No